CLINICAL TRIAL: NCT03423615
Title: Lay Fieldworker Led Comprehensive School Health Program for Rural Primary Schools in India
Brief Title: Lay Fieldworker Led School Health Program for Rural Primary Schools
Acronym: CHHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Broadleaf Health and Education Alliance (Other); Darjeeling Ladenla Road Prerna (DLRP) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-2105
Record Dates: First submitted 2018-01-20; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Health Promotion; Diarrhea
Keywords: School Health Services; Health Education; Primary Schools; Republic of India
MeSH Terms: conditions — Diarrhea; Health Education

STUDY DESIGN:
Intervention Model Description: We will use a stepped-wedge cluster controlled model to reflect the pragmatic enrollment and crossover of schools between intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHHIP Arm (Experimental): All enrolled students in schools in the CHHIP Arm were eligible to receive the CHHIP intervention. The CHHIP intervention was delivered by lay fieldworkers (SHAs). Intervention activities included:
  1. Health Education: activity-based curriculum with lessons delivered once per week. Units include hygiene, nutrition, safety, disease prevention& management, and social, emotional, and behavior development.
  2. Basic Primary Health Services: school-based treatment including deworming and iron supplementation; screening and referral programs including growth monitoring, well-child exam, vision screening, epilepsy screening, and oral health; psychosocial and counseling support for students with atypical behaviors.
  3. Health School Environment: improvements to physical infrastructure including latrines and water systems; modeling of positive behavior reinforcement, inclusive learning environment, and avoidance of corporal punishment.
  Interventions: Behavioral: Comprehensive Health & Hygiene Improvement Program (CHHIP)
- Comparison Arm (No Intervention): All enrolled students in schools in the Comparison Arm received school health activities as were routinely available in their school, through their curriculum, or through special events.

INTERVENTIONS:
Behavioral: Comprehensive Health & Hygiene Improvement Program (CHHIP) — CHHIP is an intense, multi-component holistic school health program based on the WHO Health Promoting School framework and designed for implementation by lay fieldworkers.
  Arms: CHHIP Arm

SUMMARY:
School-aged children in low and middle-income countries (LMIC) face significant challenges to their health and development which contribute to poor academic achievement. Multi-component comprehensive school health programs guided by the World Health Organization's (WHO) Health Promoting Schools (HPS) framework have been shown to positively impact health outcomes. Such programs are implemented widely throughout the world. However, in LMIC the scope and reach of school health programs are limited by human resource constraints. A key challenge to effective implementation has been the identification of effective delivery agents.

A potential alternative approach is to leverage existing community members as lay fieldworkers for the delivery of school health promotion. Our hypothesis is that lay-fieldworkers can effectively implement comprehensive school health programs in resource-constrained primary schools. This hypothesis will be tested by retrospectively analyzing data obtained during a 5-year pilot of a school health program (CHHIP) in rural primary schools of the Darjeeling Himalayas of India.

DETAILED DESCRIPTION:
The Comprehensive Health and Hygiene Improvement Program (CHHIP) is an intense multi-component comprehensive school health program. The content of the program is structured around three reinforcing components: 1) health education, 2) basic primary health services, and 3) a healthy school environment. This holistic approach is based on the WHO's Health Promoting Schools framework and designed in accordance with the Indian National Rural Health Mission's operational guidelines for the school health programme. Delivery of the program is led by lay fieldworkers termed School Health Activists (SHAs). SHAs are existing community members without formal background or certification. The SHAs serve as the primary delivery agent for all components of the program.

From 2012 to 2016, the CHHIP program was implemented by Darjeeling Prerna, an Indian non-governmental organization, in the rural Darjeeling Himalayas, a region of the state of West Bengal in India. The program was implemented in both low-cost private and government primary schools. A convenience sample of 22 primary schools (13 government and 9 low-cost private) was chosen by the project team. Program implementation occurred in 16 schools and was led by 4 lay fieldworkers. The intervention was implemented as a community development program with a rigorous evaluation component and all data was collected prospectively. This research study was added post-hoc with data transmitted to the research team prior to any analysis.

The study is designed as a mixed methods stepped-wedge cluster controlled evaluation. A primary school will be a cluster and each step in the study will be a single academic year. In accordance with guidelines for the design and evaluation of complex evaluations, this study will couple process evaluation with that of definitive impact. The intervention will be evaluated across three domains: outcomes, implementation, and mechanism of impact.

The primary impact outcome will be the incidence of diarrheal illness as assessed by 14-day parental recall. A secondary outcome, health knowledge as assessed by pre and post-test, will be utilized as a key mediator to assess for differential impact on mechanisms of impact. Statistical analysis will be carried out as a comparison between the intervention and control arms within the context of the stepped-wedge framework. The analysis will be based on individual student-level data, with the unit of assignment (schools) included as a cluster effect in the regression analysis. Exposures of interest will be explored for association with the outcome in univariate analyses. Diarrheal incidence rate ratios will be calculated via multivariable Poisson regression analysis and mean difference in health knowledge post-test scores will be obtained using a multivariable linear mixed model. All P-values will be 2-tailed and significance will be set at P<0.05.

To study implementation, process outcomes will be obtained via a series of descriptive analysis. Coverage rates for individual health interventions and performance evaluations scores expressed as means and standard deviations will be obtained. In consultation with the project team, the research study team will define benchmarks for reach and fidelity, prior to analysis of data.

Qualitative data will be integrated with quantitative data via a process of triangulation. This data was obtained from parents and teachers in focus groups and lay fieldworkers in semi-structured interviews. Coding and analysis of the qualitative data will begin with a deductive coding method. Common themes, including important contrary opinions, will be identified and illustrative quotes will be selected.

All quantitative analysis will be done in SPSS and qualitative analysis completed in CATMA. The reporting and presentation of this trial will be in accordance with the Transparent Reporting of Evaluations with Nonrandomized Designs (TREND) guidelines.

ELIGIBILITY:
Three geographic regions representative of rural Darjeeling were identified and all primary schools in these regions were considered eligible for participation in the intervention. A convenience sample of 22 schools were pragmatically selected.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2909 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Diarrhea incidence | March, July, and November of each academic school year through the duration of the study (up to 5-years)
  Diarrheal incidence was assessed by verbal parental recall based on previous 14-days.

SECONDARY OUTCOMES:
Health Knowledge | Baseline and week 32 of each academic year through the duration of the study (up to 5-years)
  Health knowledge was assessed by an internally created written health knowledge test

OTHER OUTCOMES:
Coverage rates | At the time of intervention delivery
  Coverage rates for selected health interventions will be assessed as the proportion of eligible students receiving the intervention.
Fidelity | At the time of intervention delivery
  Fidelity was assessed by performance assessment scores of SHA service delivery based on standardized rubrics.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Matergia, MD, Principal Investigator — Center for Global Health, Colorado School of Public Health, Aurora, Colorado, USA

REFERENCES:
- [Derived] Matergia M, Ferrarone P, Khan Y, Matergia DW, Giri P, Thapa S, Simoes EAF. Lay Field-worker-Led School Health Program for Primary Schools in Low- and Middle-Income Countries. Pediatrics. 2019 Apr;143(4):e20180975. doi: 10.1542/peds.2018-0975. Epub 2019 Mar 14. PMID 30872330